CLINICAL TRIAL: NCT03581201
Title: The Relationship of the Intestinal Microbiome and the Dynamic Changes of Sex Hormone Concentrations in Women at Childbearing Age
Brief Title: The Relationship of the Intestinal Microbiome and the Menstrual Cycle
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Collaborators: University of Vienna (Other)
Responsible Party: Principal Investigator, Alexandra Kautzky-Willer, Univ. Prof. Dr., Head of the Gender Medicine Unit, Medical University of Vienna
Other Study IDs: MB2018
Record Dates: First submitted 2018-06-10; First posted 2018-07-10 (Actual); Last update posted 2019-09-03 (Actual); Status verified 2019-08

CONDITIONS: Sex Hormones; Microbial Colonization
Keywords: intestinal microbiome; oral contraceptives; estrogens; bacterial population; hormone status; glucose profiles; lipid parameters; body composition
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Oral contraception: Healthy females at childbearing age with oral contraception.
  Interventions: Diagnostic Test: Laboratory measurements; Diagnostic Test: Stool samples; Diagnostic Test: Bioimpedance analysis
- No contraception: Healthy females without any contraception at all.
  Interventions: Diagnostic Test: Laboratory measurements; Diagnostic Test: Stool samples; Diagnostic Test: Bioimpedance analysis

INTERVENTIONS:
Diagnostic Test: Laboratory measurements — Laboratory measurements will be collected every week during the Duration of one menstrual cycle and includes the following:
  * Hormone analysis
  * Clinical chemistry
  * Complete blood count
  * Adipokines
  * Glucose and HbA1c-levels
  * Urinary Chemistry
Diagnostic Test: Stool samples — For a Duration of one menstrual cycle the study participants will be instructed to collect stool samples every two days. The investigation of the intestinal microbiome will be done by sequencing the 16S rRNA gene.
Diagnostic Test: Bioimpedance analysis — The Bioimpedance analysis (BIA) is used for the measurement of body composition and will be done at every study visit.

SUMMARY:
In the present study the dynamic changes of the intestinal microbiome are observed over a 4-week period in the different stages of the menstrual cycle in women at childbearing age. The focus is on how the dynamic changes of sex hormones during a menstrual cycle of women at childbearing age (with or without contraception) are related to microbiological colonization of the gut. In Addition the Expression of the β-glucuronidase by the bacteria will be investigated.

DETAILED DESCRIPTION:
Our gut has a complex and diverse bacterial population which is called the microbiome. The number of bacteria in the intestine is estimated to exceed 10^14. The composition of the microbiome is individual and changes over the lifetime of the host.

The composition of a healthy microbiome consists more than 90% of bacteria from the Bacteroidetes and Firmicutes phyla types. Nevertheless the microbiome varies even between healthy individuals and evolves over the lifetime.

Most of the microorganisms are not pathogen, thus they have been shown to interact with several physiological processes in our body. In Addition it has been shown that the bacterial population has an impact on building our gut epithelial cells, our immunology and the defence against pathogens.

Interestingly estrogen and the microbiome seem to be under reciprocal influence. In our body estrogen is only active in the deconjugated form. Therefore, after it was conjugated in the liver, the bacteria in the gut can perform a deconjugation through the secretion of the enzyme ß-glucuronidase. Ultimately, the activated estrogen is going back into blood circulation, otherwise it would leave the body through bile excretion. The composition of the microbiome is fundamental, because the presence and abundance of different gene expressions varies between the different types of bacteria. The bacterial genes which are responsible for metabolizing estrogens are called the estrobolome. However, data whether there is a relationship of the changes of the sex hormones during the menstrual cycle and the intestinal microbiome in women is sparse.

Parts of the estrogens circulating in the body are metabolised in the liver and are then secreted to the intestine conjugated with glucuronide. The intestinal microbiota could potentially affect estrogen metabolism via Beta-glucuronidase activity. Beta-glucuronidase is an enzyme that catalyses the deconjugation of estrogen. As a consequence, it may bind to estrogen receptors and unfold its downstream effects.

ELIGIBILITY:
Inclusion Criteria:

* women at childbearing age
* age 18-40 years
* BMI 18.5-24.9 kg/m²
* taking oral contraceptives
* not having any contraceptives

Exclusion Criteria:

* chronic and acute infectious diseases
* history of taking antibiotics or probiotics in the last 3 months
* gastrointestinal disorders in the last 3 months
* Polycystic Ovary Syndrome
* disorders of the menstrual cycle (e.g. oligomenorrhea, anovulation)
* other than mediterranean diet

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: In total, 20 patients (10 subjects with oral contraceptives and 10 subjects without oral contraceptives or any contraceptive at all) between 18 and 40 years and a body mass index (BMI) between 18 and 24 kg/ m² will be examined in this study.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2018-07-18 (Actual); Primary Completion 2020-06-13 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
Changes of the B-Glucuronidase, expressed by the intestinal microbiome, during the menstrual cycle in women at childbearing age | Up to 7 weeks
  Parts of the estrogens circulating in the body are metabolised in the liver and are then secreted to the intestine conjugated with glucuronide. The intestinal microbiota could potentially affect estrogen metabolism via β-glucuronidase activity. β-glucuronidase is an enzyme that catalyses the deconjugation of estrogen. As a consequence, it may bind to estrogen receptors and unfold its downstream effects.
  RNA and total DNA will be extracted from the fecal samples and microbiome community composition will be assessed by sequencing the 16s ribosomal RNA gene. Then reverse transcription of the total RNA and targeted amplification and sequencing of β-glucuronidase gene fragment will be applied in order to find out which bacteria are producing the β-glucuronidase enzyme.
  Furthermore, the enzymatic activity in the samples will be measured using the β-glucuronidase colorimetric assay with p-nitrophenol glucuronide.

SECONDARY OUTCOMES:
Changes of the Beta-Glucuronidase during the menstrual cycle in women with oral contraception | Up to 7 weeks
Changes of the Beta-Glucuronidase during the menstrual cycle in women without any contraception | Up to 7 weeks
Changes of the intestinal microbiome during the menstrual cycle in women at childbearing age with- and without contraception | Up to 7 weeks
Relationship of the β-Glucuronidase with the changes of the female sex hormones during the menstrual cycle in women at childbearing age. | Up to 7 weeks
Relationship of the intestinal microbiome with the changes of the female sex hormones during the menstrual cycle in women at childbearing age. | Up to 7 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Kautzky-Willer, Prof. Dr., Principal Investigator — Department of Internal Medicine III, Clinical Division of Endocrinology and Metabolism, Unit of Gender Medicine, Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria